CLINICAL TRIAL: NCT02912481
Title: Real-time Ultrasound-guided Arterial Catheterization in Pediatric Patients: Comparison of Success Rate Among the Arteries
Brief Title: Posterior Tibial Artery Catheterization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: H-1606-108-771
Record Dates: First submitted 2016-09-21; First posted 2016-09-23 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Arterial Catheterization

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- Posterior tibial artery (Experimental): real time ultrasound guided arterial catheterization on the posterior tibial artery
  Interventions: Procedure: posterior tibial artery
- Radial artery (Active Comparator): real time ultrasound guided arterial catheterization on the radial artery
  Interventions: Procedure: radial artery
- Dorsalis pedis artery (Active Comparator): real time ultrasound guided arterial catheterization on the dorsalis pedis artery
  Interventions: Procedure: dorsalis pedis artery

INTERVENTIONS:
Procedure: posterior tibial artery
  Arms: Posterior tibial artery
Procedure: radial artery
  Arms: Radial artery
Procedure: dorsalis pedis artery
  Arms: Dorsalis pedis artery

SUMMARY:
Arterial catheterization in small children is challenging, even for experienced anesthesiologists. For successful arterial catheterization, the arterial diameter, cross-sectional area, and depth from the skin surface are important considerations, especially in pediatric patients. THe investigators examined the posterior tibial artery (PTA) and dorsalis pedis artery (DPA) using ultrasound (US) to find a reasonable alternative arterial cannulation site to the radial artery (RA) in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing general anesthesia needing invasive arterial monitoring

Exclusion Criteria:

* Surgery involving the both hands or foots

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 275 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
first access success rate | immediate after anesthetic induction, maximum 10 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- SNUH, Seoul, Jongro Gu, South Korea